CLINICAL TRIAL: NCT04903366
Title: Absorption and Safety of Topically Applied Timolol for Treatment of Chronic Cutaneous Wounds
Brief Title: Absorption and Safety of Topical Timolol to Treat Chronic Wounds
Status: Completed | Type: Observational
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roslyn Rivkah Isseroff, M.D., Professor, Chief of Dermatology, VA Northern California Health Care System
Other Study IDs: 17-10-00798
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma, Open-Angle; Chronic Wounds
Keywords: Timolol; Catecholamine; Absorption
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Timolol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic wound: Any chronic wound, for greater than 30 days with minimal improvement
  Interventions: Drug: Timolol Maleate
- Glaucoma: Any diagnosis of glaucoma and active prescription of timolol drops
  Interventions: Drug: Timolol Maleate

INTERVENTIONS:
Drug: Timolol Maleate — timolol maleate 0.5% gel-forming solution

SUMMARY:
Topical timolol has been used primarily as eye drops to treat glaucoma for many years. Recent clinical experience has broadened its off-label use for a number of skin conditions, including slow-healing wounds. While there have been extensive safety studies performed on timolol administration to treat the eye, to date, no studies have documented absorption of timolol after applied on chronic wounds. Thus, the purpose of this study is to determine the blood levels of timolol in patients after topical administration to a chronic wound, and compare these levels with those of patients after administration of the same drug formulation on the eye for the indication of glaucoma.

DETAILED DESCRIPTION:
Chronic wounds, such as diabetic foot ulcers, venous leg ulcers and pressure ulcers are serious problems in our health system, with limited therapeutic options available to improve healing. Our laboratory and animal work has suggested that timolol, a safe medication, currently used as an eye drop for treatment of glaucoma, can heal these ulcers.

Timolol, is a nonselective, beta1/beta2 adrenergic receptor antagonist, widely used for the management of ocular hypertension or open-angle glaucoma. Most recently, there have been many case reports published that suggest that timolol can be used topically to aid in the healing of chronic, recalcitrant ulcers and wounds; however, concern over the medication's systemic effects needs to be further explored and elucidated. The systemic absorption of timolol eye drops and the medications systemic side effects have been well established; however, this has not before been examined in patients receiving topical timolol for chronic wounds. Now that this beta blocker has promising evidence for a role in the topical management of chronic wounds, the safety of this drug in topical use is of interest.

The importance of this study is in the exploration of the safety of timolol in the topical treatment of chronic wounds. If the systemic absorption from topical application to chronic wounds is found to be equivalent or less than that from ophthalmic drops, then a strong argument can be made regarding the relative safety of Timolol.

To investigate the safety profile of topical timolol application, blood levels will be measured to determine the systemic absorption of timolol. To do this, we proposed an observational cross-sectional comparative study with two groups of patients: one group receiving topical timolol for chronic wounds and the other receiving ophthalmic timolol for the management of glaucoma. Serum levels of timolol will be quantified using high performance liquid chromatography (HPLC), and the levels between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Using physician-prescribed timolol as directed
* The ability to read, understand, and sign informed consent for blood draw and release of medical information forms
* For wound group: documented chronic wound (greater than 30 days, with minimal improvement), with any type of wound.
* For glaucoma group: diagnosed with ocular hypertension or open-angle glaucoma.

Exclusion Criteria:

* Patient is not currently prescribed timolol or currently taking oral metoprolol
* History of any type of heart block
* History of bradycardia (heart-rate less than 60 beats per minute (bpm))
* History of documented hypotension
* History of asthma or chronic obstructive pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans treated at VA Northern California Health Care System from the Dermatology Wound Clinic and the Eye Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Mean plasma concentration of timolol in each group | Blood was drawn 1 hour after drug administration
  For both groups, after administration of timolol drops as prescribed, one 6 mL blood was drawn. After centrifugation, the plasma from both groups was frozen at -80°C until assay.

SECONDARY OUTCOMES:
Systemic levels of timolol dose per body weight | Blood was drawn 1 hour after drug administration
  Measurement of timolol dose per kilogram body weight plotted against the systemic plasma timolol level
Systemic levels of timolol by dose and wound type | Blood was drawn 1 hour after drug administration
  Measurement of mean plasma levels of timolol in the different wound categories (e.g., venous, diabetic, pressure ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Rivkah R Isseroff, MD, Principal Investigator — VA Northern California Health Care System
Locations (1):
- VA Northern California Health Care System, Mather, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallegos AC, Davis MJ, Tchanque-Fossuo CN, West K, Eisentrout-Melton A, Peavy TR, Dixon RW, Patel RP, Dahle SE, Isseroff RR. Absorption and Safety of Topically Applied Timolol for Treatment of Chronic Cutaneous Wounds. Adv Wound Care (New Rochelle). 2019 Nov 1;8(11):538-545. doi: 10.1089/wound.2019.0970. Epub 2019 Oct 16. PMID 31637100